CLINICAL TRIAL: NCT00193635
Title: Pilot Study of Mycophenolate Mofetil in Congenital Uropathies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Hoffmann-La Roche (Industry); University of Medicine and Dentistry of New Jersey (Other); New York Presbyterian Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL214; CEL214
Record Dates: First submitted 2005-09-09; First posted 2005-09-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Congenital Urological Abnormalities
Keywords: Congenital uropathies; Mycophenolate mofetil; GFR; Iothalamate clearance; Urine cytometry; Children; Congenital urological abnormalities which represent stuctural defects in the genitourinary system
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): oral MMF
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — oral drug administration
  Other Names: Cellcept

SUMMARY:
Congenital or hereditary structural anomalies of the genitourinary tract account for approximately half of all cases of end stage renal disease in the pediatric population. Despite optimal medical management, when the GFR falls below 50 ml/min/1.73 M2, nearly 40% of affected children will require dialysis or a renal transplant within 2 years. At present, there is no specific treatment for patients with congenital uropathies that can retard the progressive loss of kidney function and forestall the need for renal replacement therapy.

There is evidence in experimental animals and in patients with chronic renal failure (CRF) that immunoeffector mechanisms are activated within the renal parenchyma. Infiltration of the kidney by macrophages, monocytes, and lymphocytes, activation of renal tubular epithelial cells, and release of pro-inflammatory cytokines result in fibrosis and irreversible organ damage.

Mycophenolate mofetil (MMF) is a new immunosuppressive agent that is used to prevent acute rejection in kidney transplant recipients. It attenuates renal damage in the remnant kidney model of CRF in which there is no primary immunological injury. Therefore, this pilot study is designed to test the hypothesis that immunosuppressive treatment with MMF in children with structural causes of CRF will be safely tolerated and that this therapy will retard progressive decline in renal function.

Patients with congenital uropathy, 3-16 years of age and with a GFR less than 50 ml/ml/1.73 M2, will be treated with MMF for 24 months. The two primary endpoints are: (1) safety and tolerance of the drug; and (2) need for dialysis or kidney transplantation. It is anticipated that the MMF will be free of significant toxicity and that administration of the drug will reduce the frequency of progression to end stage renal disease from 38% to 19%. Patients will be followed at 3-month intervals and they will undergo serial assessment of proteinuria, estimated GFR and iothalamate clearance, urinary cytokine excretion, urine flow cytometry, and immunologic testing.

The significance of this pilot study is that it may provide evidence in support of a randomized, double-blind, placebo-controlled trial of immunological treatment of congenital structural causes of CRF in children

DETAILED DESCRIPTION:
Sustained activation of the immune system may contribute to progressive renal injury in all forms of chronic kidney disease. There is extensive proliferation of renal tubular epithelial cells and fibroblasts within the kidney of patients with chronic renal failure (CRF). The fibroblasts manifest an activated myofibroblast phenotype, evidenced by expression of alpha smooth muscle actin. This change is accompanied by infiltration of the renal interstitium with macrophages, lymphocytes, and other immunocompetent cells. The cells are also activated and release numerous cytokines and inflammatory mediators. These substances exacerbate the injury process by recruiting additional immunoeffector cells into the kidney parenchyma and stimulating the production and secretion of pro-inflammatory molecules. These findings suggest that immunosuppressive medications may be beneficial in the treatment of congenital uropathies. In fact, mycophenolate mofetil (MMF) (10-30 mg/kg/day) has been given to rats that had been subjected to a 5/6 nephrectomy. Uremia in this remnant kidney model is not the consequence of primary immunological disease. MMF treatment for 30-60 days did not prevent intraglomerular hypertension or the alterations in renal hemodynamics that characterize the adaptation to reduced renal mass. However, the extensive infiltration of the renal interstitium by proliferating lymphocytes was markedly attenuated by MMF treatment. Moreover, despite the relatively selective anti-metabolic effect of MMF on lymphocytes, there was a significant reduction in macrophage infiltration in the tubulointerstitium. This beneficial change was associated with a significant reduction in albuminuria and glomerulosclerosis after 60 days of MMF treatment. Combined treatment with the MMF and the angiotensin converting enzyme (ACE) inhibitor, lisinopril, to rats with reduced renal mass diminished tubulointerstitial infiltration by macrophages and T cells even more than MMF therapy alone and nearly normalized urinary protein excretion. Thus, pharmacological treatment with MMF attenuated the progression of "nonimmunological" renal disease in the remnant kidney model without favorably impacting on intraglomerular hemodynamics or the hypertrophic response to peptide growth factors.

MMF is a well-tolerated, safe, and effective immunosuppressive medication in adult and pediatric recipients of cadaveric and living-related renal transplants.

HYPOTHESIS AND SPECIFIC AIMS This open-label pilot study is designed to test the hypothesis that there is sustained activation of immunoeffector systems that mediate progressive loss of renal function in children with congenital uropathies. Immunosuppressive therapy can inhibit this process and retard the rate of decline in kidney function in pediatric patients with structural, non-immunological kidney conditions.

Specific Aim#1: Determine whether administration of mycophenolate mofetil (MMF) to pediatric patients with a glomerular filtration rate (GFR) <50 ml/min/m2 due to congenital uropathies such as dysplasia/hypoplasia, obstructive uropathy, and reflux nephropathy is safe and well tolerated.

Specific Aim#2: Determine whether administration of mycophenolate mofetil (MMF) diminishes the rate of progressive decline in GFR and the frequency of ESRD in pediatric patients with a glomerular filtration rate (GFR) <50 ml/min/m2 due to congenital uropathies.

RESEARCH DESIGN AND METHODS Clinical Definitions CRF: GFR <50 ml/min/1.73 m2

Congenital uropathy: One of the following categories of kidney disease:

1. Dysplasia/hypoplasia
2. Congenital obstructive uropathy: This category will include children born with structural abnormalities that are associated with renal parenchymal damage, e.g. Prune-Belly syndrome, posterior urethral valves, myelomeningocele.
3. Reflux nephropathy
4. Hereditary non-immunological tubular disorders

The threshold for CRF has been selected to enable recruitment of a sufficient number of patients into this pilot study in a timely fashion. In addition, at this stage in the disease course, renal function can be expected to decline during a relatively short follow-up period. Patients with this degree of CRF have nearly a 40% chance of requiring dialysis or a transplant within 2 years. This will increase the possibility of demonstrating a therapeutic benefit secondary to treatment with MMF. The diagnosis of the congenital urological disease will be established based upon appropriate use of radiological imaging tests and, if necessary, surgical procedures.

Inclusion criteria:

1. Age: 3-16 years
2. Congenital uropathy
3. Presence of CRF

The lower age limit will enable enrollment of children who are reasonably cooperative, are able to take a liquid MMF preparation orally twice a day, and in whom an iothalamate clearance can be performed without requiring bladder catheterization. The upper limit on age will enable all of the subjects to complete the 2-year study protocol prior to 18 years of age, the standard cut-off for enrollment into pediatric clinical trials.

Exclusion criteria:

1. Diagnosed primary hepatic, hematological, or immunological disease such as HIV infection that may increase the potential risks of MMF
2. Known sensitivity to MMF
3. Glomerular disease defined on clinical or histopathological grounds

The rate of decline in estimated GFR during the 6 months prior to entry into the study will be recorded in all patients. However, this value will not serve as an exclusion criterion. Even patients with evidence of rapid decline in GFR, i.e. >25% in the previous 6 months, will be eligible. Such a rapid deterioration is unlikely to occur in the children with congenital uropathy who are enrolled in this pilot study, based on the natural history of this form of kidney disease.

Sample Population It is anticipated that 12 patients will be enrolled at approximately 4 centers in this multicenter open-label pilot study of MMF in children with CRF due to congenital uropathies.

Proposed Intervention with MMF All patients will be treated with MMF in this open-label pilot study. Study Phases

There will be two phases in this open-label pilot study:

1. RUN-IN (2 months): Informed consent will be obtained from parents of eligible patients before beginning this phase of the study. Assent will be obtained according to IRB regulations at each participating center.

   During the 2-month Run-In period, eligible patients will be taken off all medications that are contraindicated by the protocol (see below, Adjunctive Treatments). At the discretion of the attending pediatric nephrologist, children may be placed on an ACE inhibitor drug. The dose must be stabilized 4 weeks prior to the onset of the Treatment Period.
2. TREATMENT (24 months): GFR will be measured by iothalamate clearance at the start of and at the end of the 12-month Treatment Period. Patients whose estimated GFR is <50 ml/min/1.73 M2 during the Run-in Period will be included regardless of the GFR determination using the iothalamate clearance at the beginning of the Treatment Period. This will reflect the prevailing clinical practice in which GFR is routinely determined using formula estimates rather than more precise clearance methods. HIV testing will be done at the first visit of the Treatment Period and MMF treatment will not be commenced until the HIV-negative status of each eligible patient is confirmed.

MMF Dosing The target therapeutic dosage of MMF will be 600 mg/m2 body surface area/dose, maximum dose 1 g, given orally twice a day. MMF will be started at 200 mg/m2 BID and increased at biweekly intervals. The full treatment dose, 600 mg/m2 BID, will be achieved at 4 weeks.

Safety parameters The dose will be adjusted downward by 200 mg/m2/BID if a child develops gastrointestinal complaints, anemia (hematocrit <25%), or an absolute neutrophil count (ANC) 1,000-1,500. If after 1 week GI toxicity continues or any of the laboratory studies remain abnormal, the dose will be further reduced in decrements of 200 mg/m2/BID. If any of these problems persist subsequently, the drug will be stopped. In a case of severe toxicity, more rapid reduction of MMF is allowed at the attending pediatric nephrologist's discretion. If ANC is less than 1000, the drug will be stopped. The need to discontinue MMF treatment in more than 20% of the study patients will be considered an unacceptable high frequency of MMF intolerance in this pilot trial.

Adjunctive treatments The use of ACE inhibitors will not be contraindicated in patients who are enrolled in this study. However, these agents must be started prior to enrollment into the trial and the initial dose will not be increased during the remainder of the 2-year study protocol. Administration of recombinant human growth hormone to children who enroll in this pilot study will be permitted if the attending pediatric nephrologist has already prescribed it. In addition, patients may receive erythropoietin to treat anemia and to prevent the need for red blood cell transfusions.

Supplemental doses of antioxidants such as vitamin E will be contraindicated for study participants. In addition, patients in this trial will not be give any other immunosuppressive therapy. All other treatments will be left to the discretion of the attending pediatric nephrologist.

Clinical Assessment

Pre-enrollment, interval and final visits:

CLINICAL: BP, urine protein:creatinine ratio (Upr/c), microalbuminuria (Ualb/cr), iothalamate clearance IMMUNOLOGICAL: HIV testing at the initial visit. NUTRITION: Counseling to provide RDA for protein and 125% RDA for calories

All serum and urine samples will be stored at -70 degrees C after analysis for future testing if new clinical research findings indicate the value of performing a novel assay to assess disease progression in children with congenital uropathies.

Frequency of interval assessment Run-in Period: Monthly x 2 Treatment Period: Monthly x 3 Then every 3 months for duration of study

Primary Endpoints

1. Safety of MMF in children with congenital uropathies
2. Frequency of ESRD in children with congenital uropathies

Anticipated findings It is predicted that MMF will be well tolerated by at least 80% (10 out of 12) of the children with a congenital uropathy and a GFR <50 ml/min/1.73m2. It is also anticipated that MMF will reduce the incidence of ESRD by 50% and, thus, at most 2 out of 12 patients treated with MMF in this protocol will require dialysis or transplant.

Timeline of pilot study It is anticipated that it will take 3 months to set up an Administrative Center at Schneider Children Hospital, design Clinical Reporting Forms, and create a database at a Data Coordinating Center. Patients would be recruited over the next 3 months. In order to complete a 2-year Treatment Period, the entire study would last for 3½ years.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-16 GFR <50 ml/min/1.73 m2 Congenital abnormality of urinary tract

Exclusion Criteria:

* Known hepatic, hematologic, GII, infectious disease Sensitivity to MMF Glomerular disease

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2002-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Reduction in GFR | 24 month treatment period

SECONDARY OUTCOMES:
Safety and tolerance of MMF | 24 month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — Schneider Children's Hospital of North Shore-LIJ Health System
Locations (3):
- United States (3):
  - Robert Wood Johnson Medical center, New Brunswick, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - Cornell Weill Medical Center, New York, New York

REFERENCES:
- [Derived] Trachtman H, Christen E, Frank R, Rini J, Palestro C, Perelstein E, Weiss L, Tarapore F, Fortune S, Horowitz J. Pilot study of mycophenolate mofetil for treatment of kidney disease due to congenital urinary tract disorders in children. Am J Kidney Dis. 2008 Oct;52(4):706-15. doi: 10.1053/j.ajkd.2008.03.035. Epub 2008 Jun 13. PMID 18554762